CLINICAL TRIAL: NCT06849518
Title: Study of Longitudinal Plasma PD-L1 Testing With Immunotherapy in Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ballad Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2276376
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: A Circulogene liquid biopsy testing for plasma NGS ctDNA and plasma cfRNA PD-L1 expression will be drawn (i) pre-treatment, (ii) at cycle 2 treatment, (iii) every other cycle while on combined doublet chemotherapy-immune treatment, (iv) at 3 months post-starting treatment, (v) at 6 months post-starting treatment, and (vi) upon discontinuation of ICI treatment due to planned completed duration of ICI treatment or upon progressing disease. ICI treatment and radiographic evaluations will be standard of care as determined by the treating oncologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plasma NGS ctDNA and plasma cfRNA PD-L1 expression (Other)
  Interventions: Diagnostic Test: Circulogene liquid biopsy testing

INTERVENTIONS:
Diagnostic Test: Circulogene liquid biopsy testing — A Circulogene liquid biopsy testing for plasma NGS ctDNA and plasma cfRNA PD-L1 expression.

SUMMARY:
This is a prospective pilot study to assess dynamic changes of plasma cell-free RNA (cfRNA) PD-L1 expression in patients with lung cancer undergoing immune checkpoint inhibitor (ICI) based therapy. Results will be correlated with radiographic assessment of immunotherapy treatment response and plasma NGS ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a diagnosis of stage IV or inoperable stage IIIB NSCLC without planned primary radiation therapy undergoing anti-PD-1/L1 based ICI treatment.
2. Chemo-immune or dual anti-PD-1/L1 with anti-CTLA-4 based regimens are eligible as long as receiving an anti-PD-1/L1 monoclonal antibody.
3. A documented informed consent will be obtained prior to inclusion in the study. All discussions with patients will be held in strictest confidence and out of earshot of the general public. Patients will be fully informed that their participation in the study is voluntary. Patients may decline to be part of the study. Their decision to participate in the study will not affect the care they receive.

Exclusion Criteria:

1. No anti-PD-1/L1 monoclonal antibody treatment.
2. Planned primary radiation therapy.
3. Small-cell lung cancer histology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of plasma cfRNA PD-L1 by qPCR expression* with ICI treatment and response. | up to 24 months
  Circulogene ImmunoClear Assay

SECONDARY OUTCOMES:
Correlation of plasma cfRNA PD-L1 expression* results with any available tissue PD-L1 protein expression. | up to 24 months
  Circulogene ImmunoClear Assay

CONTACTS AND LOCATIONS:
Locations (1):
- Ballad Health Cancer Care, Kingsport, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No